CLINICAL TRIAL: NCT06483477
Title: Dermatitis During Adjuvant Irradiation for BREAst Cancer: Grade ≥2 Radiation Dermatitis in Breast Cancer Patients with or Without a Mobile Application (Reminder-App)
Brief Title: Dermatitis During Adjuvant Irradiation for BREAst Cancer:
Acronym: DAI-BREAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Southern Denmark (Other); Medical School Hamburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DAI-BREAC
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Female
Keywords: Breast cancer; Radiotherapy; Dermatitis; Mobile application
MeSH Terms: conditions — Breast Neoplasms; Dermatitis

STUDY DESIGN:
Intervention Model Description: multinational, randomized, active-controlled, parallel-group, multicenter trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Standard skin care supported by a reminder app
  Interventions: Other: Standard skin care; Device: Reminder App
- Arm B (Active Comparator): Standard skin care alone
  Interventions: Other: Standard skin care

INTERVENTIONS:
Other: Standard skin care — From the start of radiotherapy, standard skin care has to be performed by the patient. This may vary at the participating centers. At the site in Lübeck, it includes fatty cream with 2-10% urea (fatty cream alone, if patients do not tolerate urea) and, in case of pruritus, addition of mometasone furoate cream. In case of grade ≥2 moist desquamation or grade ≥3 radiation dermatitis, each day antiseptic agents will be administered for wound cleansing followed by administration of silicon or calcium alginate bandage. This treatment will be continued until moist desquamation radiation disappears and radiation dermatitis improves to grade 2. Fatty cream with 2-10% urea is applied to the irradiated skin four times daily. Mometasone furoate cream: In addition to the fatty cream with 2-10% urea, mometasone furoate cream (solution 0.1%) is applied to the irradiated skin once daily.
Device: Reminder App — In addition to standard skin care, patients are supported by a Reminder App. The purpose of the app is to remind the patients in an intuitive, unobtrusive and supportive way to perform skin care. By default, patients are reminded four times a day, but they will also be able to define a notification schedule that best suits their personal needs. The patients may postpone each required care procedure for up to 2 hours. With each procedure, the patients are guided through the skin care with simple and self-explanatory illustrations. To increase the patients' motivation, they will additionally earn points for regular and punctual performed care procedures. The patients receive a hand-out including instructions how to properly perform skin care, but they can also find an information page within the application that includes similar instructions.
  Arms: Arm A

SUMMARY:
In the randomized DAI-BREAC trial, a reminder app will be prospectively tested that reminds breast cancer patients four times each day to perform the required skin care. This will likely contribute to the reduction of grade ≥2 radiation dermatitis in these patients. A total of 268 patients will be randomized to receive standard skin care supported by a reminder app (Arm A) or standard skin care alone (Arm B). Stratification will be done using the three factors treatment volume, radiation boost, and at least one risk factor of dermatitis. Secondary aims include pain (radiation fields), patient satisfaction with the reminder app (Arm A only), impact of the app on the use of health technology (Arm A only), and benefit from support by staff members of the treating Department of Radiation Oncology and/or the UKSH academy regarding the use of the app (Arm A only).

DETAILED DESCRIPTION:
The main goal of this trial is to evaluate whether standard skin care supported by a reminder app is superior to standard skin care alone with respect to prevention of grade ≥2 radiation dermatitis in patients receiving adjuvant radiotherapy for invasive breast cancer. Radiation dermatitis will be assessed by an observer (specially trained nurse, technician, or physician) different from the person who performs the routine visit of the patient ("blinded observer concept"), at the start of radiotherapy and weekly during the course of radiotherapy, and at the end of the radiotherapy course (=EOT) according to CTCAE v5.0. Secondary aims include pain (radiation fields), patient satisfaction with the reminder app (Arm A), impact of the reminder app on the use of health technology (Arm A), and benefit from support by staff members and/or the UKSH academy regarding the use of the reminder app (Arm A).

This is a multinational, randomized, active-controlled, open-label, multicenter, parallel-group trial, which compares the following treatments of radiation related skin toxicity in patients with breast cancer: Standard skin care supported by a reminder app (Arm A) vs. standard skin care alone (Arm B). Stratification will be done using the following prognostic factors:

1. Treatment volume: Breast or chest wall alone vs. breast or chest wall plus lymph nodes
2. Radiation boost: Yes vs. no
3. At least one risk factor of dermatitis: Yes vs. no Risk factors include chronic inflammatory disease, significant cardiovascular disease, and smoking history of >10 pack years.

After registration, patients will be randomized in a 1:1 ratio to Arm A or Arm B for treatment of radiation related skin toxicity. A stratified block-randomization with random block size will be performed via electronic CRF. The results of the randomization will be visible only after the input of the stratification factors and only for the corresponding patient.

This document will be kept at the institution which performs the randomization until the end of the study. Afterwards, the original randomization list will be kept in the trial master file at the trial center of the coordinating investigator for a minimum of 10 years after the final report. The randomization will be performed via electronic CRF centrally by an external company using its standard software. The proceeding for randomization is based on standard operating procedures (SOPs) of this company. Once the randomization is allocated to the patient it cannot be changed.

In all patients, radiotherapy will be administered using hypo-fractionation with 40 Gy in 15 fractions of 2.667 Gy given on 5 days per week (overall treatment time = 3 weeks; day of 15th fraction = EOT), preferably with intensity-modulated radiotherapy (IMRT) or volumetric-modulated arc therapy (VMAT). Patients aged ≤50 years receive a sequential radiation boost to the tumor bed of 10 Gy in 5 fractions of 2.0 Gy (on 5 days per week) following whole-breast irradiation, resulting in an overall treatment time of 4 weeks (day of 20th fraction = EOT). This accounts also for patients aged ≥51 years with risk factors for local recurrence. Patients may receive concurrent systemic agents as part of their standard anticancer treatment, regardless of the participation in this trial. These agents may include tamoxifen, aromatase inhibitors, or capecitabine [10]. The systemic agents will be indicated and prescribed by treating medical oncologists or gynecologists outside this trial. Regarding dose, type and duration of treatment, contraindications, side effects, pharmacological characteristics and pharmaceutical details of these agents, please see the corresponding product information.

Standard Skin Care alone (Arm B):

From the start of radiotherapy, standard skin care has to be performed by the patient. This may vary at the participating centers. At the site in Lübeck, it includes fatty cream with 2-10% urea (fatty cream alone, if patients do not tolerate urea) and, in case of pruritus, addition of mometasone furoate cream. In case of grade ≥2 moist desquamation or grade ≥3 radiation dermatitis, each day antiseptic agents will be administered for wound cleansing followed by administration of silicon or calcium alginate bandage. This treatment will be continued until moist desquamation radiation disappears and radiation dermatitis improves to grade 2. Fatty cream with 2-10% urea is applied to the irradiated skin four times daily. Mometasone furoate cream: In addition to the fatty cream with 2-10% urea, mometasone furoate cream (solution 0.1%) is applied to the irradiated skin once daily.

Patients of Arm B will be informed about the importance of skin care prior to the start of radiotherapy and reminded during their radiotherapy course, when regularly seen by a radiation oncologist (maximum once a week).

Standard Skin Care plus Reminder App (Arm A):

From the start of radiotherapy, standard skin care has to be performed by the patient as described for Arm B. In addition, patients of Arm A are supported by a Reminder App, which is developed by the professional company Nextlabel OHG from Lübeck. The purpose of the app is to remind the patients in an intuitive, unobtrusive and supportive way to perform skin care. By default, patients are reminded four times a day, but they will also be able to define a notification schedule that best suits their personal needs.

Questionnaire regarding the Reminder App and its impact on the use of health technology:

At the end of their radiotherapy course (= EOT), the patients of Arm A will be asked to complete a questionnaire regarding their satisfaction with the Reminder App. In case of a dissatisfaction rate >20%, the reminder app is considered to require modifications before it can be used in future studies. In case of a dissatisfaction rate >40%, it will be considered not useful. This questionnaire also includes questions regarding the impact of the app on the use of health technology. Elderly patients aged ≥65 years will be compared to younger patients aged <65 years to identify potential differences between both age groups and the need for support regarding the use of the reminder app.

Sample size calculation

The primary goal of this randomized trial is to evaluate whether standard skin care supported by a reminder app is superior to standard skin care alone with respect to preventing grade ≥2 radiation dermatitis during adjuvant hypo-fractionated radiotherapy for breast cancer. According to sample size calculations, 131 patients are required per study arm within the Full Analysis Set. Considering that 2% of patients will not qualify for Full Analysis Set, a total of 268 patients should be randomized. The following analysis sets will be defined for this trial:

Safety Analysis Set: All randomized participants who started radiotherapy. Full Analysis Set: All randomized patients who have started either therapy with arm A or with arm B and provide any data on the primary endpoint. The Full Analysis Set will be analyzed according to the Intention-to-Treat principle, i.e. patients will be analyzed in their initial group of randomization.

Per Protocol Set: All patients of the Full Analysis Set excluding patients if any of the following criteria are met:

* Administration of less than 75% of the planned radiation dose if the reason for discontinuation was any other than death or unacceptable toxicity
* More than 50% missing data on the primary study endpoint All patients in the Per Protocol Set will be analyzed within their group of actual treatment received.

Statistical analyses:

All data recorded in the electronic case report forms describing the study population and toxicity will be analyzed descriptively. Categorical data will be presented in contingency tables with frequencies, percentages and their 95% confidence intervals. Continuous data will be summarized with at least the following: frequency (n), median, quartiles, mean, standard deviation (standard error), minimum and maximum. Number of patients with protocol deviations during the study and listings describing the deviations will be provided.

In general, chi-square tests will be used to compare percentages in a two-by-two contingency table, replaced by Fisher´s exact test if the expected frequency in at least one cell of the associated table is less than 5. Stratified two-by-two contingency tables will be analyzed using Cochran-Mantel-Haenszel tests. Logistic regression models serve as multivariable methods for binary endpoint data. Comparison of ordinal variables between treatment arms will be performed using the asymptotic Wilcoxon-Mann-Whitney test, replaced by its exact version in case of ordinal categories with small number of categories and/or sparse data within categories. Any shift in location of quantitative variables between study groups will be performed with the Wilcoxon-Mann-Whitney tests as well.

Time-to-event data will be analyzed by Kaplan-Meier methods, when merely non-informative censoring occurs. For statistical comparison, the log rank-test will be provided supplemented by multivariate Cox proportional hazards models.

The data analysis will be performed according to the statistical analysis plan (SAP), and which will be finalized prior to database lock and prior to any statistical analysis.

To evaluate the rate of patients experiencing grade ≥2 radiation dermatitis during their course of radiotherapy, the worst documented grade during radiotherapy and at EOT is considered, even if patients have missing visits or discontinue radiotherapy prematurely. This reflects the "treatment policy estimand" approach.

The rate of patients experiencing grade ≥2 radiation dermatitis will be statistically compared using the Cochran-Mantel-Haenszel Chi-square test on a two-sided significance level of 5%. This test is the natural non-parametric extension of the Chi-square test for testing the treatment effect, while adjusting for the effects of the stratification variables used for randomization. In case of uneven distribution to stratification groups, which may result in very small groups the strata might be pooled for analysis. The decision to pool strata for the analysis will be made before data base lock and before the final analysis of the data.

For further assessment of the robustness of the results, a logistic regression model for grade ≥2 radiation dermatitis will be applied including the parameters used for stratification. A model including additional patient characteristics will be fitted for exploratory purposes. The confirmatory evaluation will be performed within the Full Analysis Set; the Per Protocol Set serves for further sensitivity analyses.

The visual analogue scale pain prior to radiotherapy, during radiotherapy and at EOT will be subjected to descriptive analyses. pain potential differences in pain between treatment arms, the scores will be subjected to descriptive analysis. For graphical visualization Box-Whisker diagrams will be provided. Moreover, the change from baseline values will be considered and subjected to descriptive analyses. Friedman tests and Wilcoxon-Mann Whitney tests may be applied for comparison of study visits.

At the EOT-visit, patient satisfaction with the reminder app in arm A will be evaluated and subjected to standard statistical methods. In case of a dissatisfaction rate >20%, the reminder app needs modifications. In case of a dissatisfaction rate >40%, it will be considered not useful. In addition, the questions on the impact of the app on the use of health technology will be evaluated descriptively. Elderly patients aged ≥65 years will be compared to younger patients aged <65 years to identify potential differences between both age groups and the need for support regarding the use of the reminder app. Standard statistical tests serve as a tool for exploratory comparison of age groups.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven invasive breast cancer
2. Indication for adjuvant hypo-fractionated radiotherapy
3. Possession of and ability to use a smartphone
4. Female gender
5. Age ≥18 years
6. Written informed consent
7. Capacity of the patient to contract

Exclusion Criteria:

1. Pregnancy, Lactation
2. Expected non-compliance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of grade ≥2 radiation dermatitis | through study completion, an average of 4 weeks
  Radiation dermatitis will be assessed according to CTCAE v5.0.

SECONDARY OUTCOMES:
Pain score | through study completion, an average of 4 weeks
  Pain (skin within radiation fields) will be assessed with a visual analogue scale (self-assessment, ranging from 0 = no pain to 10 = maximum pain). Furthermore, the intake of analgesics will be documented.
Rate of patient satisfaction with the reminder app | through study completion, an average of 4 weeks
  Patient satisfaction with the reminder app will be assessed with a specific questionnaire (Arm A only).
Degree of the impact of the reminder app | through study completion, an average of 4 weeks
  Impact of the reminder app on the use of health technology will be assessed with a specific questionnaire (Arm A only).
Rate of patient satisfaction with support | through study completion, an average of 4 weeks
  4. Benefit from support by staff members of the treating Department of Radiation Oncology and/or the UKSH academy regarding the use of the reminder app will be assessed with a specific questionnaire (Arm A only).

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Rades, MD, FASTRO, Principal Investigator — Dept. of Radiation Oncology, University of Lubeck, Germany
Locations (5):
- Vejle Hospital, University Hospital of Southern Denmark, Vejle, Southern Denmark, Denmark
- Germany (4):
  - Medical Practice for Radiotherapy and Radiation Oncology, Hanover, Lower Saxony
  - Medical School Hamburg, Schwerin Campus, Schwerin, Mecklenburg-Vorpommern
  - Malteser Hospital St. Franziskus, Flensburg, Schleswig-Holstein
  - Department of Radiation Oncology, University of Lübeck and University Medical Center Schleswig-Holstein, Lübeck

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rades D, Narvaez-Wolf CA, Dziggel L, Staackmann C, Radtke M, Timke C, Kristiansen C, Duma MN, Yu NY, Janssen S. Dermatitis during adjuvant irradiation for breast cancer (DAI-BREAC): a randomized controlled trial investigating whether grade >/=2 dermatitis during radiotherapy for breast cancer can be reduced by a mobile application that reminds patients to perform skin care. Trials. 2025 Mar 20;26(1):99. doi: 10.1186/s13063-025-08800-2. PMID 40114285